CLINICAL TRIAL: NCT02030834
Title: Phase IIa Study of Redirected Autologous T Cells Engineered to Contain Anti-CD19 Attached to TCRz and 4-Signaling Domains in Patients With Chemotherapy Relapsed or Refractory CD19+ Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 13413, 818607
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2020-10

CONDITIONS: Non-Hodgkins Lymphoma (NHL) Patients, With CD19+B Cell Lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): murine CART19
  Interventions: Biological: CART-19
- Cohort B (Experimental): T cell/histiocyte-rich Diffuse Large B Cell Lymphoma (DLBCL) treated with murine CART19
  Interventions: Biological: CART-19
- Cohort C (Experimental): Diffuse Large B Cell Lymphoma (DLBCL) treated with humanized CART19
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — Single infusion of CART-19 cells administered by i.v. injection (total dose of 1 - 5 x108 CART-19 cells, calculated as a range of 2-50% transduced cells in total cells).

SUMMARY:
Phase IIa study to estimate the efficacy of a single infusion of autologous T cells expressing CD19 chimeric antigen receptors expressing tandem TCR and 4-1BB (TCR /4-1BB) costimulatory domains (referred to as CART-19 or CTL019 cells) in non-Hodgkins Lymphoma (NHL) patients. The duration of active protocol intervention is approximately 24 months from screening visit. The protocol will require approximately 48 months to complete.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects with CD19+ B cell lymphomas with no available curative treatment options (such as autologous or allogeneic SCT) who have a limited prognosis (several months to <2 year survival) with currently available therapies will be enrolled. The study will enroll 51 evaluable subjects as follows:
* CD19+ Lymphoma

Cohort A Subjects:

a. Follicular lymphoma, previously identified as CD19+ i. At least 2 prior chemotherapy or immunochemotherapy regimens (not including single agent monoclonal antibody therapy) ii. Patients who progress within 2 years after second or higher line of therapy will be eligible. For instance, patients who have progression of lymphoma < 2 years after second or greater line therapy, but who have responded to their most recent treatment (3rd line or higher) will be eligible. Patients may have progression, stable disease or responding disease at the time of enrollment.

iii. Patients with a history of large cell transformation are eligible. b. Mantle cell lymphoma, previously identified as CD19+ i. Beyond 1st CR with relapsed disease, progressive disease during first line rituximab-chemotherapy combination, or persistent disease after first line rituximab-chemotherapy combination and not eligible or appropriate for conventional allogeneic or autologous SCT.

ii. Relapsed after prior autologous SCT. c. Diffuse large B cell lymphoma, previously identified as CD19+ i. Residual disease after primary therapy and not eligible for autologous SCT ii. Relapsed or persistent disease after prior autologous SCT iii. Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT iv. Patients with an antecedent history of follicular lymphoma or CLL/SLL are eligible.

Cohort B Subjects:

a. Diffuse large B cell lymphoma, previously identified as CD19+ CD19 i. Residual disease after primary therapy and not eligible for autologous SCT ii. Relapsed or persistent disease after prior autologous SCT iii. Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT iv. Patients with an antecedent history of follicular lymphoma or CLL/SLL are eligible.

v. Patients with T cell/histiocyte-rich disease as confirmed by surgical pathology report

Cohort C Subjects:

a. Diffuse large B cell lymphoma, previously identified as CD19+ i. Residual disease after primary therapy and not eligible for autologous SCT ii. Relapsed or persistent disease after prior autologous SCT iii. Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT iv. Patients with an antecedent history of follicular lymphoma or CLL/SLL are eligible.

* Age ≥18 years
* Creatinine < 1.6 mg/dL
* ALT/AST < 3x upper limit of normal
* Bilirubin <2.0 mg/dL, unless subject has Gilbert's Syndrome (<3.0 mg/dL)
* Any relapse after prior autologous SCT will make patient eligible regardless of other prior therapy.
* Patients with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and:

  1. Have no active GVHD and require no immunosuppression
  2. Are more than 6 months from transplant
* Measurable or assessable disease according to the "Revised Response Criteria for Malignant Lymphoma" (Cheson et al., J. Clin. Onc., 1999)108. Patients in complete remission with no evidence of disease are not eligible.
* Performance status (ECOG) 0 or 1.
* Left Ventricle Ejection Fraction (LVEF) > 40% confirmed by ECHO/MUGA
* Written informed consent is given. Successful T cell test expansion (first 10 subjects).

Exclusion Criteria

* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum pregnancy test at enrollment. A urine pregnancy test will be performed within 48 hours before infusion.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary. For additional details regarding use of steroids
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification (see Appendix 1).
* HIV infection.
* Patients with active CNS involvement by malignancy. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment
* Patients in complete remission with no assessable disease.
* Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schuster, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Schuster SJ, Svoboda J, Chong EA, Nasta SD, Mato AR, Anak O, Brogdon JL, Pruteanu-Malinici I, Bhoj V, Landsburg D, Wasik M, Levine BL, Lacey SF, Melenhorst JJ, Porter DL, June CH. Chimeric Antigen Receptor T Cells in Refractory B-Cell Lymphomas. N Engl J Med. 2017 Dec 28;377(26):2545-2554. doi: 10.1056/NEJMoa1708566. Epub 2017 Dec 10. PMID 29226764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 50 | 3 | 10
Completed | 39 | 3 | 7
Not Completed | 11 | 0 | 3
Not completed — Death | 4 | 0 | 0
Not completed — Manufacturing failure | 2 | 0 | 1
Not completed — Disease progression | 2 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lack of funding | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 50 | 3 | 10 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 2 | 8 | 47
  >=65 years | 13 | 1 | 2 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 1 | 2 | 23
  Male | 30 | 2 | 8 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 48 | 3 | 9 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Overall Response (i.e. Either Complete Response or Partial Response) Evaluated at Three Months Post Infusion.
Description: Responders will include those patients achieving complete response (CR), complete response unconfirmed (CRu) and partial response (PR) using anatomic imaging such as CT or MRI to assess tumor volume or, in the event of bone marrow involvement, morphologic and immunohistochemical confirmation that the bone marrow infiltrate has been cleared.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 39 | 3 | 7
Participants | 24 | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 5/50 | 0/3 | 2/10
Serious Adverse Events (participants affected / at risk) | 32/50 | 3/3 | 5/10
Other Adverse Events (participants affected / at risk) | 39/50 | 3/3 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=50) | Cohort B (N=3) | Cohort C (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0 — Scotoma left eye
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 — Incarcerated umbilical hernia
Fever (General disorders) | 6 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 20 | 2 | 4
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — Influenza A
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — Streptococcal Bacteremia
Lung infection (Infections and infestations) | 3 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Second primary cancer
Encephalopathy (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=50) | Cohort B (N=3) | Cohort C (N=10)
Anemia (Blood and lymphatic system disorders) | 14 | 1 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 | 0 — Splenomegaly
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 8 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0 — Fogginess
Flashing lights (Eye disorders) | 0 | 0 | 1
Floaters (Eye disorders) | 1 | 0 | 0
Optic nerve disorder (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 0
Constipation (Gastrointestinal disorders) | 9 | 1 | 1
Diarrhea (Blood and lymphatic system disorders) | 8 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 — Barrett's Esophagus
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 2 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1 | 1
Chills (General disorders) | 0 | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0 — White on tongue
Edema limbs (Gastrointestinal disorders) | 8 | 1 | 1
Edema trunk (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 23 | 2 | 3
Fever (General disorders) | 5 | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 | 0 — Rigors
Localized edema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 0
Pain (General disorders) | 7 | 1 | 2
Allergic reaction (Immune system disorders) | 2 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 3 | 0 | 0
Gum infection (Infections and infestations) | 2 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 0 — Giardia in stool
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — Bronchiolitis
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — Clostridium difficile
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — flu
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — Lymphadenitis: inguinal
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — Upper Respiratory Infection
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 — UTI
Lung infection (Infections and infestations) | 2 | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 1
Skin infection (Infections and infestations) | 3 | 0 | 0
Small intestine infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 10 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Head Laceration
Alanine aminotransferase increased (Investigations) | 11 | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 3 | 3
Blood bilirubin increased (Investigations) | 6 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 2 | 0 | 0
Cholesterol high (Investigations) | 2 | 0 | 0
Creatinine increased (Investigations) | 6 | 1 | 1
Fibrinogen decreased (Investigations) | 0 | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 1 — Headache
Lymphocyte count decreased (Investigations) | 7 | 0 | 2
Lymphocyte count increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 19 | 2 | 5
Platelet count decreased (Investigations) | 10 | 2 | 1
Weight gain (Investigations) | 2 | 0 | 0
Weight loss (Investigations) | 4 | 0 | 0
White blood cell decreased (Investigations) | 13 | 1 | 3
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 3 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 13 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 18 | 2 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 12 | 2 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Body aches in joints and muscles
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Calcium Pyrophosphate Deposition Disease
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 — Cramps
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Lateral epicondylitis
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Muscular atrophy
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 — Labral tear
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Twitching: finger
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Basal cell carcinoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Melanoma (T1A)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Squamous cell carcinoma
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 11 | 1 | 3
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Movements involuntary (Nervous system disorders) | 1 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 — Tingling
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Spasticity (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 3 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 2 | 0 | 0
Hallucinations (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 — Hydroureteronephrosis
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 — Urinary hesitancy
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 — Urine: foamy
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Lungs: decreased breath sounds
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Lungs: crackles
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Morning cough and sputum production
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Actinic keratosis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Bloody lips
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Contact dermatitis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 — Erythematous rash
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Night sweats
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 — Rash
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Skin excoriation
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Verruca vulgaris
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 — Warts
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Vescular rash
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Folliculitis
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 4 | 0 | 0
Hypotension (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 2 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0 — Fluid overload
Vascular disorders - Other, specify (Vascular disorders) | 1 | 1 | 1 — Night sweats
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0 — Livedo reticularis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02030834/Prot_SAP_000.pdf